CLINICAL TRIAL: NCT04046692
Title: Cross - Observational Study About Hospital School Experience for the Reduction of Distress, Pain and Negative Experience and for the Promotion of School Experience's Continuity. the Point of View of Teachers, Children and Parents
Brief Title: School Activity for the Reduction of Distress, Pain and Negative Emotions in Children Experiencing Hospital School
Status: Completed | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Collaborators: University of Florence (Other)
Responsible Party: Principal Investigator, Rosanna Martin, Principal Investigator, Meyer Children's Hospital IRCCS
Other Study IDs: Hospital_School
Record Dates: First submitted 2019-07-29; First posted 2019-08-06 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-10

CONDITIONS: Hospital School Experience
Keywords: hospital school; pain; distress; negative emotions; school continuity; child
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- children in hospital school in contact with outside school: children experience school's lesson with the hospital teacher in the school's room or into their bedrooms and the investigator give before/after the lesson 2 questionnaire (PANAS-C and PH-C) and the VAS to evaluate the aim's study. Then, the investigator asks the children to make 2 paintings: one about the hospital school experience (what is for him/her the hospital school) and one about the outside school (what he/she do/did outside during school).
  Interventions: Other: Hospital School Experience, point of view of the children
- children in hospital school NOT in contact with outside school: it's the same of the previous group ("children experiencing hospital school still in contact with outside school"); the only difference of this group is that children are not in contact with the outside school.
  Interventions: Other: Hospital School Experience, point of view of the children
- hospital teachers: teachers have to answer to some questions (qualitative interview) and fill in CEESQ schedule
  Interventions: Other: Hospital School Experience, point of view of the hospital teachers
- outside teachers: teachers have to answer to some questions (qualitative interview) and fill in CEESQ schedule
  Interventions: Other: Hospital School Experience, point of view of the non hospital teachers
- Parents: parents have to answer some questions (qualitative interview)
  Interventions: Other: Hospital School Experience, point of view of parents

INTERVENTIONS:
Other: Hospital School Experience, point of view of the children — Operators of the PANAS-C, PH-C and VAS ask the children to answer the questionnaire before/after the school lesson; then they ask the children to make 2 paintings about hospital and not hospital school experience.
  Groups: children in hospital school NOT in contact with outside school; children in hospital school in contact with outside school
Other: Hospital School Experience, point of view of the hospital teachers — operators interview hospital teachers and make them complete a questionnaire (CEESQ)
  Groups: hospital teachers
Other: Hospital School Experience, point of view of the non hospital teachers — operators interview the teachers and make them complete a questionnaire (CEESQ)
  Groups: outside teachers
Other: Hospital School Experience, point of view of parents — Operators interview parents
  Groups: Parents

SUMMARY:
Aim of present study is to evaluate the efficacy of hospital school experience in the reduction of distress, pain and negative emotion in children from 8 to 12 years old, hospitalized in oncology and pediatric wards. Investigators also want to explore the ideas and opinions of teachers and parents about hospital school service.

Hypothesis: the investigators expect a reduction in pain, distress and negative emotions.

DETAILED DESCRIPTION:
The school service into the hospital was born as an attempt to support emotionally, relationally and cognitively the hospitalized children, who have to spend a lot of time alone, without being educated by teachers with their classmates. There are not many studies in the Italian contest about this issue and with the present study the investigators intended to implement the acknowledgement about this theme.

The principal aim of this study is to explore if the school service reduces negative emotions experienced by oncological children as well as perceived pain and distress. To evaluate this aims, the investigators organized the study in 3 sections: the first is about the emotions experienced by oncological children between 8 and 12 years old, who benefit from the school service into the hospital; the second is about their parents' opinions and believes about the hospital school service; the third is about opinions, training and educational method dedicated by hospital school teachers and not hospital school teachers (who previously thought to our oncology children sample).

ELIGIBILITY:
Inclusion Criteria for children:

* age between 8 and 12 years old
* knowledge of Italian language
* consent for study participation
* recovery
* be/not be in contact with classmates (group A and group B)

Exclusion Criteria for Children:

* patients who have already had hospital school experience in the past
* cognitive disability
* patients that cannot complete the study because of health or mental issues incoming during the period of the research

Inclusion criteria for hospital teachers:

* Italian knowledge
* Being a hospital teacher

Exclusion criteria for hospital teachers:

- Have earlier experience as a hospital children in other hospitals

Inclusion criteria for not hospital teachers:

* Italian knowledge
* Being a teacher of the hospitalized children in the past or present time exclusion criteria for not hospital teachers:
* A past experience as a hospital teacher

Inclusion criteria for parents:

* Italian knowledge
* consent for study participation
* Health or mental issues that can cause problems in completing questionnaires or answering questions

Exclusion criteria for parents:

* Cognitive disability
* Health or mental issues that can cause problems in completing questionnaires or answering questions

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children 8-12 years old in oncology and pediatric wards, having hospital school into Meyer Hospital; parents of these children; hospital and not hospital teachers of the patients included in the study
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Change in Positive and Negative affect before/after hospital school experience | PANAS - C is completed by the child before and after the school experience (average 3 months); it takes around 5 minutes for each investigation.
  PANAS - C (Positive and Negative Affect Scale for Children): original version by Laurent (1999), italian version by Ciucci and collaborators. 30-item numerical scale assessing two dimensions (positive and negative affect, 15-item each) on a 5 point likert scale. Validated for children between 8 and 12 years old. Aim of this scale is to evaluate the presence of positive and negative emotions before/after an experience/activity.
Change in Distress level before/after hospital school experience | PH - C is completed by the child before and after the school experience (average 3 months); it takes around 3 minutes for each investigation.
  PH - C (Psychological Hyperarousal Scale for Children): original version by Laurent (2004), italian version by Ciucci and collaborators. Numerical scale composed by 18 items measured on a 5 point Likert Scale. Aim of this scale is to evaluate the presence/absence of distress before and after the activity.
Change in Pain level before/after hospital school experience | VAS is completed by the child before and after the school experience (average 3 months); it takes around 30 seconds for each investigation.
  visual analogue scale (VAS) for children, by Scott, Ansell, & Huskisson (1977). It's a likert scale measuring perceived pain from 0 (no pain) to 10 (maximum pain).

SECONDARY OUTCOMES:
explorative interview for parents | Investigators interview the parent in a silent and private room within 1 year after child's recruiting
  it's a partially structured interview concerning ideas and opinions of parents about hospital school service
explorative interview for hospital teachers | investigators interview the hospital teacher in a silent and private room within 3 months after child's recruiting
  it's a partially structured interview concerning ideas and opinions of hospital teachers about hospital school service, methods of learning and teaching
explorative interview for outside teachers | investigators arranged an appointment to interview the teacher within 1 year after child's recruiting
  it's a partially structured interview concerning ideas and opinions of outside teachers about hospital school service
research form for investigator | within 3 months after child's recruiting, the researcher observes a lesson and then fills in the form
  it's a research partially structured form regarding informations about how it's organised hospital school service
research form for the outside teacher | through study completion, an average of 1 year, the outside teacher fill in the form after a lesson
  it's a research partially structured form regarding informations about how it's organised hospital school service
child's emotions and ideas about hospital school service | within 1 year after child's recruiting, investigators ask the child to draw when present in the Oncology Day Hospital or in the oncology/pediatric ward and then pick the draw
  investigators ask the child to draw the hospital school service and then is asked what he/she has drawn, what it represents, what's for him/her the best moment of hospital school
child's emotions and ideas about outside school service | within 1 year after child's recruiting, investigators ask the child to draw when present in the Oncology Day Hospital or in the oncology/pediatric ward and then pick the draw
  investigators ask the child to draw the outside school service and then is asked what he has drawn, what it represents, what's for him/her the best moment of school; also, children is asked if he/she perceives a difference between outside school and hospital school service
emotions and self efficacy of hospital teachers | the investigator asks the teacher to fill in the questionnaire, within 3 months after child's recruiting
  CEESQ (Crèche Educators Emotional Style Questionnaire): italian version by Ciucci, Baroncelli and Toselli (2015); numerical scale measuring emotions and self efficacy on a likert scale from 0 to 5; it takes around 10/15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Rosanna Martin, MSc, Study Director — Meyer Children's Hospital IRCCS
Locations (1):
- Meyer Chidren's Hospital, Florence, Firenze, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Decision has to be shared between Meyer Children's Hospital, University of Florence and Clinical Trial Office of Meyer Hospital

REFERENCES:
- [Background] Antonelli E, Vagnoli L, Ciucci E, Vernucci C, Lachi F, Messeri A. A Comparison of Nonpharmacologic Interventions on the Emotional State of Children in the Emergency Department. Pediatr Emerg Care. 2019 Feb;35(2):81-88. doi: 10.1097/PEC.0000000000000900. PMID 27749803
- [Background] Charlton A, Larcombe IJ, Meller ST, Morris Jones PH, Mott MG, Potton MW, Tranmer MD, Walker JJ. Absence from school related to cancer and other chronic conditions. Arch Dis Child. 1991 Oct;66(10):1217-22. doi: 10.1136/adc.66.10.1217. PMID 1953006
- [Background] Clatworthy S, Simon K, Tiedeman ME. Child drawing: hospital--an instrument designed to measure the emotional status of hospitalized school-aged children. J Pediatr Nurs. 1999 Feb;14(1):2-9. doi: 10.1016/S0882-5963(99)80054-2. PMID 10063243
- [Background] Clatworthy S, Simon K, Tiedeman M. Child drawing: hospital manual. J Pediatr Nurs. 1999 Feb;14(1):10-8. doi: 10.1016/S0882-5963(99)80055-4. No abstract available. PMID 10063244
- [Background] Georgiadi, M., & Kourkoutas, E. E. (2010). Supporting pupils with cancer on their return to school: a case study report of a reintegration program. Procedia-Social and Behavioral Sciences, 5, 1288-1282.
- [Background] Hughes AA, Kendall PC. Psychometric properties of the Positive and Negative Affect Scale for Children (PANAS-C) in children with anxiety disorders. Child Psychiatry Hum Dev. 2009 Sep;40(3):343-52. doi: 10.1007/s10578-009-0130-4. Epub 2009 Jan 14. PMID 19142724
- [Background] Katz LF, Leary A, Breiger D, Friedman D. Pediatric cancer and the quality of children's dyadic peer interactions. J Pediatr Psychol. 2011 Mar;36(2):237-47. doi: 10.1093/jpepsy/jsq050. Epub 2010 Jun 2. PMID 20522423
- [Background] Laurent J, Catanzaro SJ, Joiner TE Jr. Development and preliminary validation of the physiological hyperarousal scale for children. Psychol Assess. 2004 Dec;16(4):373-80. doi: 10.1037/1040-3590.16.4.373. PMID 15584796
- [Background] Pelander T, Lehtonen K, Leino-Kilpi H. Children in the hospital: elements of quality in drawings. J Pediatr Nurs. 2007 Aug;22(4):333-41. doi: 10.1016/j.pedn.2007.06.004. PMID 17645961
- [Background] af Sandeberg M, Johansson E, Bjork O, Wettergren L. Health-related quality of life relates to school attendance in children on treatment for cancer. J Pediatr Oncol Nurs. 2008 Sep-Oct;25(5):265-74. doi: 10.1177/1043454208321119. Epub 2008 Jul 22. PMID 18648091
- [Background] Worchel-Prevatt, F. F., Heffer, R. W., Prevatt, B. C., Miner, J., Young-Saleme, T., Horgan, D., ... & Frankel, L. (1998). A school reentry program for chronically ill children. Journal of school psychology, 36(3), 261-289.
- [Background] Yilmaz MC, Sari HY, Cetingul N, Kantar M, Erermis S, Aksoylar S. Determination of school-related problems in children treated for cancer. J Sch Nurs. 2014 Oct;30(5):376-84. doi: 10.1177/1059840513506942. Epub 2013 Sep 27. PMID 24076657